CLINICAL TRIAL: NCT06036186
Title: Early Feasibility, Randomized Crossover and Double-Blind Design, Study for the Treatment of Heart Failure With Preserved Ejection Fraction (HFpEF) Associated With Hypertension Utilizing Right Atrial Pacing Regulated by the PressurePace™ System (RelieveHFpEF-II)
Brief Title: Study for the Treatment of Heart Failure With Preserved Ejection Fraction Associated With High Blood Pressure Using Right Atrial Pacing Controlled by the PressurePaceTM System
Acronym: RelieveHFpEFII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BaroPace Inc. (Industry)
Collaborators: JSS Medical Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: BP011
Record Dates: First submitted 2023-08-16; First posted 2023-09-13 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2023-09

CONDITIONS: Heart Failure With Preserved Ejection Fraction (HFpEF); Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BaroPacing treatment (Experimental): Group 1 will use BaroPacing for the first 3 weeks (day 8 to day 28) and then switch to standard treatment for another 3 weeks (day 29 to day 49).
  Interventions: Device: BaroPacing treatment
- Standard treatment (Active Comparator): Group 2 will use standard treatment for the first 3 weeks (day 8 to day 28) and then switch to BaroPacing for another 3 weeks (day 29 to day 49).
  Interventions: Device: Standard treatment

INTERVENTIONS:
Device: BaroPacing treatment — BaroPacing for the first 3 weeks (day 8 to day 28) and then crossover to standard treatment for another 3 weeks (day 29 to day 49).
  Arms: BaroPacing treatment
Device: Standard treatment — Individual Standard treatment as prescribed by the Physician to each subject for the first 3 weeks (day 8 to day 28) and then crossover to BaroPacing for another 3 weeks (day 29 to day 49).
  Arms: Standard treatment

SUMMARY:
This study is a prospective, double blind, self-controlled, randomized, cross-over study to evaluate the feasibility, efficacy, and safety of treating patients with Heart Failure with preserved Ejection Fraction (HFpEF) associated with hypertension using the PressurePace™ system of Right Atrial Pacing regulated by blood pressure in subjects with dual chamber pacemakers.

The objective of this study is to show that blood pressure-controlled right atrial pacing improves exercise tolerance, improves heart failure symptoms, and improves hypertension control in subjects with HFpEF associated with hypertension compared to conventional bradycardia pacing alone.

DETAILED DESCRIPTION:
This study is a prospective, double blind, self-controlled, randomized, cross-over study to evaluate the feasibility, efficacy, and safety of treating patients with Heart Failure with preserved Ejection Fraction (HFpEF) associated with hypertension using the PressurePace™ system of Right Atrial Pacing regulated by blood pressure in subjects with dual chamber pacemakers. No surgery, intervention or implant will occur during this study. All subjects enrolled in the study already have a dual chamber pacemaker implanted for standard clinical indications.

The objective of this study is to show that blood pressure-controlled right atrial pacing improves exercise tolerance, improves heart failure symptoms and improves hypertension control in subjects with HFpEF associated with hypertension compared to conventional bradycardia pacing alone.

Each subject will have an office/clinic visit. Once the subject signs informed consent, the pacemaker will be interrogated by trained personnel. If all the inclusion/exclusion criteria are met, then the pacemaker will be connected to the pacemaker manufacturer's interrogation module which will be connected to the BaroPace interface. The system will run with clinical oversight in the office to determine suitability for outpatient function and subject usability. The system will then be used by the subjects for the duration of the study always with the direct supervision of a trained Clinical Research Coordinators.

Subjects that met all inclusion and exclusion criteria will be entered into the baseline phase (Day 1 to Day 7) where subjects will continue to receive their baseline antihypertensive medications while on standard baseline pacing parameters. Subjects will have at baseline screening day and day 7, 24-hour Ambulatory BP monitoring (ABPM). On Screening Day subjects will undergo a 2 D echo to assess ejection fraction, 6-Minute Walk test and a treadmill using the Modified Bruce Protocol on screening and Day 7. On Day 7, if subject has >3 lbs. weight loss, or >10 mmHg drop in SBP or >5 mmHg drop in DBP (mean of the past 3 12-hour BP readings at home) or is unable to tolerate at least 3 minutes on the Modified Bruce Protocol treadmill, or walk at least 225 meters during the 6-Minute Walk test, the subject will be discontinued from the study. Subjects that continue in the study will be randomized into two groups (8 subjects in each group), group 1 will use BaroPacing for the first 3 weeks (day 8 to day 28) and then switch to standard treatment for another 3 weeks (day 29 to day 49). Group 2 will use standard treatment for the first 3 weeks (day 8 to day 28) and then switch to BaroPacing for another 3 weeks (day 29 to day 49). Total study duration for a subject will be 7 weeks (49 +/- 5 days).

At the end of 49 days, the subject will return to the office/clinic, the external system components will be disconnected, and the subject's pacemaker will be returned to pre-study parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Have a Pacetronix dual chamber pacemaker implanted for > 2 weeks that is more than 6 months from ERI (elective replacement indicator).
2. Ages: Adult subjects > 35 years and < 90 of age.
3. Have heart failure with preserved ejection fraction defined as ejection fraction > 45 percent.
4. Have hypertension (SBP >135 mmHg) within 30 days before the start of screening, despite at least one or more medication for the treatment of hypertension.
5. Screening average right atrial pacing < 50% and average intrinsic/pacing heart rate < 70 bpm over the previous clinical monitoring period of the pacemaker diagnostics of at least 14 days
6. Blood pressure of no less than 135 systolic and a diastolic blood pressure no less than 85 mm Hg at initial screening over 3 readings in 30 minutes in the sitting position, in the left arm.
7. Able to tolerate at least 3 minutes of a Modified Bruce Protocol Treadmill
8. Physically capable and willing to perform repeated 6-minute walk tests associated with the study, and a baseline distance of at least 225 meters. Symptoms limiting the duration of the 6-minute walk test must be due to heart failure alone.
9. Willing and able to sign consent.
10. Stable medications for Hypertension for at least 4 weeks prior to screening.

Exclusion Criteria:

1. A resting SBP > 170 mmHg, or < 130 SBP at screening average over 3 readings in 30 minutes. The readings will be taken with the blood pressure cuff on the subject's left arm while seated after at least ten minutes of rest. Consecutive readings will be taken at least 10 minutes apart.
2. A resting DBP > 120 mmHg, or < 80 at screening average over 3 measurements in 30 minutes.
3. Physical or psychological condition which would impair study participation.
4. End Stage Renal Disease on haemodialysis
5. Indications for emergency surgery at time of screening or planned surgery before the 49-day follow-up
6. Pregnant or breast-feeding.
7. Hospitalized in the prior six months for a heart attack, stroke, or TIA, or have a history of blood-pressure related syncope in last 6 months.
8. Have a pacemaker that is currently the subject of a manufacturer's recall or regulatory advisory of malfunction.
9. Prone to atrial or ventricular arrhythmias with altered pacing.
10. Unstable from a cardiovascular standpoint, such as on-going chest pain, the diagnosis of heart failure with reduced EF, or who report being ill or otherwise uncomfortable, medically, or psychologically at the time of study.
11. Unable to interact and execute commands with the BaroPace modules during the screening phase.
12. Taking short acting Nifedipine or Clonidine or taking ISA Beta Blockers; Acebutolol, Pindolol, Sectral or Visken

Ages: 35 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-08-26 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-04-12 (Actual)

PRIMARY OUTCOMES:
Modified Bruce Protocol treadmill total exercise time | At Screening Day, Day 7, Day 28, Day 49
Absence of Related Serious Adverse events | From screening to end of study- Day 49

SECONDARY OUTCOMES:
NYHA class position | At Screening Day, Day 7, Day 28 and Day 49
Change from baseline of the total distance in 6 minutes | At Screening Day, Day 7, Day 28, Day 49
  The change from baseline on the 7th day of the total distance in 6 minutes, in meters, that the patient can walk compared to 6 minutes walked on day 28 and 49. Baseline will be compared to both treatment and control. The 6-minute walk test will be performed according to the American Thoracic Society guidelines.
Changes in The Minnesota Living with Heart Failure Questionnaire administered | At Screening Day, Day 7, Day 28, Day 49
  The Minnesota Living with Heart Failure Questionnaire is a quality-of-life questionnaire. At every 12-hour interval during the study the subject will be asked on the computer tablet a few questions, asking how much you're the treatment has affected the enrolled subject's life on a scale of 0, 1, 2, 3, 4 or 5. Zero denoting no adverse affect on life and 5 denoting very much adverse affect on life.
Quality of life questions for measuring changes in sense of well-being during intervals of perceived changes in RA pacing | Every 12 hours throughout the 21 day treatment duration.
  It is a 3 point scale, Better=2, same=1 worse=0 reduction of Afib: How many episodes in a 21 day period.
Systolic blood pressure change from baseline | after 21 days or less of treatment
  At least 5 mmHg drop in systolic blood pressure change from baseline
Proportion of subjects with a Systolic blood pressure drop | at the end of 21 days
  Proportion of subjects with a SBP drop >= 5 mmHg
Duration of response of Systolic blood pressure after lowering | at the end of 21 days
  Duration of response of SBP after lowering >= 5 mmHg
Drop in diastolic blood pressure change from baseline | after 21 days or less of treatment
  At least 3 mmHg drop in diastolic blood pressure change from baseline
Proportion of subjects with a diastolic blood pressure drop | at the end of 21 days
  Proportion of subjects with a DBP drop >= 3 mmHg
Duration of response of diastolic blood pressure after lowering | at the end of 21 days
  Duration of response of DBP after lowering >= 3 mmHg
Reduction in the number of antihypertensive medications | at the end of 21 days
  Reduction in the number of antihypertensive medications or a reduction in milligrams of one or more medications
Reduction in atrial fibrillation | every 12 hour visit on screening, first 7 days, randomization to 21-day period, in final 21 days, for total of 7 weeks
  Reduction in atrial fibrillation monitored by telemetry and downloaded to PressurePace™
Rate of intolerance to increases in right atrial pacing | every 12 hour visit on screening, first 7 days, randomization to 21-day period, in final 21 days, for total of 7 weeks
  Rate of intolerance to increases in right atrial pacing requiring reduction to a prior lower level of right atrial pacing

OTHER OUTCOMES:
Feasibility of real-time closed loop programming of a pacemaker atrial rate based on controlled algorithm. | every 12 hour visit on screening, first 7 days, randomization to 21-day period, and in final 21 days, for total of 7 weeks
  real time programming worked=1, did not work=0
Feasibility of subject's real-time subjective inputs as a moderator of pacemaker atrial rate function and PressurePace™ | every 12 hour visit on screening, first 7 days, randomization to 21-day period, and in final 21 days, for total of 7 weeks
  real-time inputs resulted in moderating pacemaker atrial rate worked=1, did not =0
Real-time closed-loop performance of commands to regulate atrial rate pacing parameters. | every 12 hour visit on screening, first 7 days, randomization to 21-day period, and in final 21 days, for total of 7 weeks
  worked=1, did not work=0
Subject's report of changes in sense of well-being during intervals of increased right atrial pacing. | every 12 hour visit on screening, first 7 days, randomization to 21-day period, and in final 21 days, for total of 7 weeks
  Reported no change=1, reported change to un-well =0
Subjective inputs by the subject on how he/she is feeling | every 12 hour visit on screening, first 7 days, randomization to 21-day period, and in final 21 days, for total of 7 weeks
  Reported yes=1 reported no=0

CONTACTS AND LOCATIONS:
Locations (3):
- India (3):
  - Maharaja Agrasen Superspeciality Hospital, Clinical Research Department, Basement, Main Building, Room No-09, Sector-07, Agrasen Aspatal Marg, Central Spine, Vidyadhar Nagar,, Jaipur, Rajasthan
  - Dr. C. M. Chopra Hospital & Heart Care Centre, Jaipur, Rajasthan
  - L.P.S. Institute of Cardiology, G.S.V.M Medical College, Kanpur, Uttar Pradesh

IPD SHARING:
Plan to Share IPD: No